CLINICAL TRIAL: NCT01534169
Title: Function of Regulatory T Cells Improved by Treatment With an Intrathyroid Injection of Dexamethasone in Graves' Patients
Brief Title: Function of Regulatory T Cells Improved by Dexamethasone in Graves' Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiao-Ming Mao (Other)
Responsible Party: Sponsor-Investigator, Xiao-Ming Mao, Professor, MD., Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HDJP-H200829
Record Dates: First submitted 2012-02-09; First posted 2012-02-16 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Graves' Disease
Keywords: Graves' disease; Dexamethasone; Function of regulatory T cells; The proportion of Th1 and Th2 cells
MeSH Terms: conditions — Graves Disease | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Isotonic Na chloride (Experimental): The treatment strategy is the same with intervention, only the drug (dexamethasone) will be changed to isotonic Na chloride.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — The course of treatment will be last for 3 months. The intrathyroid injection of dexamethasone will be performed using a 25-gauge (0.25-mm) needle under ultrasound guidance. The injection will be performed in both lobes of the thyroid. The dosage of dexamethasone is 5mg (1.0 ml) in each lobe, twice a week during the first month of the treatment. The treatment strategy will be changed to once a week in the second month and twice a month in the third month; the dosage of dexamethasone is the same as in the first month.
  Other Names: Hexadecadrol

SUMMARY:
Antithyroid drugs is the first choice treatment of Graves' disease in China and Europe. However,the relapse rate is very high (40-60%) after therapy withdrawal, and many patients need further treatment. In our previous study, a new treatment strategy for GD has been introduced. After methimazole (18 months) combined with intrathyroid injection of dexamethasone (DEX) (3 months) treatment, the relapse rate of hyperthyroidism was markedly reduced compared with methimazole treatment alone (7.4% versus 51%) during the 2-year follow-up period. The results have been published in the 'J Clin Endocrinol Metab, 2009,94:4984-4991'. However, the mechanism by which the DEX reduces the relapse rate of GD is not fully understood. In vitro study, we have proven that DEX could effectively improve the function of regulatory T (Treg) cells and set up a new balance of T helper 1(Th1)/Th2 in GD patients(this results have been in press in the Eur J Endocrinol). In order to elucidate mechanism of this treatment strategy in vivo, we plan to recruit 20-30 patients with GD and treat those patients by intrathyroid injection of DEX combined with methimazole, and the function of Treg cells and balance of Th1/Th2 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* GD patients will have been trated with methimazole and serum levels of TSH and FT4 should be in the normal range.

Exclusion Criteria:

* Pregnancy
* Allergy to antithyroid drugs (ATD)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels more than two times the upper normal range
* Patients with coexistent endocrine or organ-specific autoimmune diseases (such as those with atopic dermatitis or bronchial asthma)
* Patients taking medications that could affect the immune system (such as corticosteroids), noncompliance because of psychiatric or other serious diseases
* Unwillingness to participate in the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Function of Regulatory T Cells | From baseline to 90 days
  Function of Treg cells will be analyzed by the proliferation rate of CD4+CD25- T cells, according to the following formula: cell proliferation rate (%) = proliferation rate of CD4+CD25- T cells co-cultured with CD4+CD25+T cells/proliferation rate of CD4+CD25- T cells alone×100%.

SECONDARY OUTCOMES:
The proportion of Th1 and Th2 cells | From baseline to 90 days
  Th1 and Th2 cells will be identified by flow cytometry analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Ming Mao, MD., Study Chair — Nanjing First Hospital Affiliated to Nanjing Medical University
Locations (1):
- Nanjing First Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Mao XM, Li HQ, Li Q, Li DM, Xie XJ, Yin GP, Zhang P, Xu XH, Wu JD, Chen SW, Wang SK. Prevention of relapse of Graves' disease by treatment with an intrathyroid injection of dexamethasone. J Clin Endocrinol Metab. 2009 Dec;94(12):4984-91. doi: 10.1210/jc.2009-1252. Epub 2009 Oct 22. PMID 19850691
- [Result] Hu Y, Tian W, Zhang LL, Liu H, Yin GP, He BS, Mao XM. Function of regulatory T-cells improved by dexamethasone in Graves' disease. Eur J Endocrinol. 2012 Apr;166(4):641-6. doi: 10.1530/EJE-11-0879. Epub 2012 Jan 4. PMID 22219499